CLINICAL TRIAL: NCT02946372
Title: Transposition of Internal Limiting Membrane in the Treatment of Macular Holes. A Descriptive Pilot Study
Brief Title: Evaluation of a New Surgical Technique for Macular Hole Which Was Not Closed After a Previous Surgery
Acronym: ILMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHRMSA 872; 2016-A01431-50 (Registry Identifier: ID/RCB)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2017-08

CONDITIONS: Retinal Perforations
Keywords: retina surgery; macula; macular hole; internal limiting membrane (ILM); vitrectomy; autologous transplantation
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ILMT (Experimental): internal limiting membrane autologous transplantation (ILMT)
  Interventions: Procedure: internal limiting membrane transplantation (ILMT)

INTERVENTIONS:
Procedure: internal limiting membrane transplantation (ILMT) — internal limiting membrane autologous transplantation (ILMT)

SUMMARY:
Macular hole is an infrequent retinal pathology (2 to 4/1000) which most often affects people aged over 60, and twice common in women than men.

The vast majority of cases are idiopathic. Without treatment, the macular hole evolves through a series of stages until the extension of the diameter (up to 500 microns and higher values). With a fully developed macular hole, patients complain of metamorphopsia and decreased visual acuity.

This pathology has clearly benefited from advances in microsurgery and better understanding of its pathophysiology. Macular hole treatment has evolved to include small-gauge pars plana vitrectomy with or without internal limiting membrane (ILM) peeling and placement of intraocular gas tamponade.

The postoperative closure rate is close to 80%, but strongly depends on the initial characteristics of the hole, its diameter remaining the main prognostic factor. Thus for macular holes <400 microns, the closure rate is close to 92% dropping to 56% for macular holes above 400 microns. In case of surgical failure, one or more reoperations can be proposed, but with a lower closure rate.

The quest for a surgical technique presenting a greater success rate is a common goal to all retinologists.

Here the investigators propose a new surgical technique, derived from the FLAP method, and consisting of an inner limiting membrane transposition.

The objective of this study is to evaluate the feasibility of a new surgical technique for the treatment of macular holes already operated but without macular hole closure, allowing these patients a new therapeutic alternative. The success of this technique will be confirmed by detecting postoperatively the presence of the transposed internal limiting membrane into the foveal region.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged over 18,
2. Patient who already received at least a macular hole surgery,
3. Period of at least 4 months since last macular hole surgery,
4. Patient who underwent peeling of the internal limiting membrane,
5. Presents in OCT an open criteria macular hole,
6. The presence of a cataract in the preoperative clinical examination is not against indication. Its removal can be integrated to the surgery,
7. Patient who signed the consent form

Exclusion Criteria:

1. Patient with against-indication or surgical anesthetic,
2. Macular Hole "flat open" or closed,
3. No progressive macular pathology other than the presence of a macular hole (retinal detachment, Macular degeneration related to age) Idiopathic and secondary macular holes are eligible if they have already been operated with the prior internal limiting membrane coat.
4. Patient unaffiliated or not the beneficiary of a social security system, or equivalent health insurance,
5. Pregnant or breastfeeding women,
6. Absence of patient consent,
7. Patient in exclusion period involved in another study,
8. Patient on administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Presence of the internal limiting membrane transposed into foveal region | 8 weeks after surgery

SECONDARY OUTCOMES:
The size and appearance of the macular hole will be assessed by optical coherence tomography (OCT) | 8 weeks after surgery
Visual acuity will be assessed by clinical examination | 8 weeks after surgery
The patient's visual comfort will be assessed using the NEI-VFQ-25 Quality of Life questionary | 8 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick LENOBLE, MD, Principal Investigator — Groupe Hospitalier de la Region de Mulhouse et Sud Alsace
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No